CLINICAL TRIAL: NCT06762990
Title: Evaluating Changes of Spino-pelvic Radiological Parameters During Muslim Prayer Positions: a Cross-sectional Study
Brief Title: Evaluating Changes of Spino-pelvic Radiological Parameters During Muslim Prayer Positions
Status: Enrolling by invitation | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmed A. Khalifa, MD, FRCS, MSc, Assistant Professor, South Valley University
Other Study IDs: 04-2024-300511
Record Dates: First submitted 2024-12-15; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Spinopelvic Relatiohship; Spinopelvic Parameters Change During Praying Positions
Keywords: spinopelvic relationship; pelvic incidence; pelvic tilt; sacral slope; lumbar lordosis
MeSH Terms: conditions — Lordosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: Plain radiographs — Plain radiographs, including the lumbar spine, pelvis, and the upper half of both femora, will be obtained using the lowest radiation dose possible. The radiographs will be obtained in five positions representing the Muslim Prayers positions, namely 1-standing, 2-Sitting in 90 degrees (both 1 and 2 are the standard positions obtained in all previous studies), 3-bowing (Ruku), 4-prostration (sujud), and 5-sitting with knees bent (Tashahud).

SUMMARY:
This observational study aims to investigate the spinopelvic relationship parameters change during the five main positions during Muslim prayers. The main questions the study is going to answer: What are the changes of the spinopelvic parameters during different Muslim prayer positions?

DETAILED DESCRIPTION:
The spinopelvic relationship refers to the intricate and dynamic interaction between the spine and the pelvis, which plays a crucial role in maintaining posture, balance, and overall musculoskeletal function. The alignment and movement of the spine and pelvis are interdependent, with changes in one structure often influencing the other. Understanding this relationship is essential for diagnosing, managing, and treating various spinal and pelvic conditions; furthermore, these parameters profoundly affect acetabular cup positioning and could affect dislocation rate after total hip arthroplasty.

Evaluating the normal spinopelvic parameters for any particular population is the first step toward detecting abnormal relationships, these were evaluated in various populations, such as Indian, Brazilian, Korean, and Caucasians.

Besides the deficiency of such reports from our area (Middle East), most of the published reports evaluated the change in spinopelvic relationship by evaluating the differences occurring from standing to 90 degrees sitting positions, which ignores most of the positions occurring during Muslim prayer, which necessitates more flexion of the hips and spine during specific position such as prostration (sujud). Activities that involve dynamic movements, such as Muslim prayer positions, can influence spinopelvic parameters. The sequence of postures in Muslim prayers, which includes standing, bowing, and kneeling, places unique demands on the spinopelvic alignment. Understanding how these positions affect spinopelvic parameters is essential for providing insights into the potential implications for musculoskeletal health, particularly in populations that engage in these activities regularly; furthermore, the possibility of proceeding with prayers after THA surgery if the dislocation risk due to impingement is low. What are the changes of the spinopelvic parameters during different Muslim prayer positions and if these changes are different between males and females and if these parameters are affected by participants' body habits, mainly the Body Mass Index (BMI).

ELIGIBILITY:
Inclusion Criteria:

Adult participants (18 to 55 years old) who are willing to volunteer to participate in the study, reporting performing prayer positions without difficulty, had no hip or spine surgeries or complaints (pain or stiffness)

Exclusion Criteria:

* Participants refusing to volunteer.
* Participants who are not able to perform prayer positions comfortably.
* Those who had prior spine or hip surgeries.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers who are working at our hospital or visiting the out patient clinic who are willing to participate to the study without any consequences after explaining for them the purpose and any harms of the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change of the spinopelvic parameters measured in spinopelvic lateral plain radiographs (in degrees) Across Five Muslims Prayer Positions | 4 months
  Spine and pelvis lateral plain radiographs will be obtained in five positions representing the Muslim Prayers positions, namely 1-standing, 2-Sitting at 90 degrees, 3-bowing (Ruku), 4-prostration (sujud), and 5-sitting with knees bent (Tashahud). The following parameters: Pelvic Incidence (PI), Pelvic Tilt (PT), Sacral Slope (SS), Lumbar Lordosis (LL), and pelvic femoral angle (PFA) will be measured in degrees by two of the authors using the Surgimap application.
  Then, Spinopelvic movements will be calculated as the difference between the standing and the remaining four positions (ΔX = ΔX (4 positions) - ΔX standing) for each of the measured spinopelvic parameters (LL, SS, PI, PT, PFA). The change in each parameter between these positions will be analyzed to understand pelvic orientation variations during prayer movements.

SECONDARY OUTCOMES:
Differences between males and females regarding the spinopelvic parameters measured in spinopelvic lateral plain radiographs (in degrees) Across Five Muslims Prayer Positions | 4 months
  Spine and pelvis lateral plain radiographs will be obtained in five positions representing the Muslim Prayers positions, namely 1-standing, 2-Sitting at 90 degrees, 3-bowing (Ruku), 4-prostration (sujud), and 5-sitting with knees bent (Tashahud). The following parameters: Pelvic Incidence (PI), Pelvic Tilt (PT), Sacral Slope (SS), Lumbar Lordosis (LL), and pelvic femoral angle (PFA) will be measured in degrees using the Surgimap application, the five parameters will be compared between males and females. Then, Spinopelvic movements will be calculated as the difference between the standing and the remaining four positions (ΔX = ΔX (4 positions) - ΔX standing) for each of the measured spinopelvic parameters (LL, SS, PI, PT, PFA), and the change in each parameter will be compared between males and females to understand the gender differences related to pelvic orientation variations during prayer movements.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. Abdelaal, MD, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No